CLINICAL TRIAL: NCT01725425
Title: The Impact of Portion Size of Foods on Mood in Normal Weight Adults 18-35
Brief Title: The Effect of Portion Sizes on Mood
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Professor, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 8964B
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Mood; Eating Patterns
Keywords: snack food (chips); fruit (red grapes) consumed in each condition; mood

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (Experimental): Participants will receive equal amounts of foods.
  Interventions: Other: Control
- Increase Portion Size (Experimental): Participants will receive increased portion sizes.
  Interventions: Other: Increase Portion Size
- Decrease Portion Sizes (Experimental): Participants will receive decreased portion sizes.
  Interventions: Other: Decrease Portion Size
- Mixed Portion Sizes (Experimental): Participants will receive mixed portion sizes.
  Interventions: Other: Mixed Portions

INTERVENTIONS:
Other: Control — The control is designed to determine average mood.
  Arms: Control
Other: Increase Portion Size — The purpose is to determine whether a change in mood will occur.
  Arms: Increase Portion Size
Other: Decrease Portion Size — The purpose is to determine whether a change in mood will occur.
  Arms: Decrease Portion Sizes
Other: Mixed Portions — The purpose is to determine if a change in mood will occur.
  Arms: Mixed Portion Sizes

SUMMARY:
The purpose of this study is to investigate whether different portion sizes will effect overall mood.

DETAILED DESCRIPTION:
The objective of this investigation is to determine whether participants will have a change in mood based on the portion size of foods served. The specific aims of the study are:

1. Determine the effect of increasing portion sizes on mood.
2. Determine the effect of decreasing portion sizes on mood.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35
* have a body mass index of 18.5 and 24.9 kg/m^2
* be an unrestrained eater( scoring less than 12 on the Three Factor Eating Questionnaire)
* Report Being a non-smoker

Exclusion Criteria:

* currently pregnant or nursing
* report being an athlete in training
* currently taking any medications that affect appetite or food intake
* Have a medical condition affecting eating or are currently following a therapeutic diet
* Report disliking foods used in the investigation
* Report having allergies to foods used in the investigation

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2012-10 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Total grams of snack food consumed | 1 year
  The snack food consumed in this investigation is Lays Potato Chips (Frito-Lay Inc., Plano, TX). Participants will be provided 50 or 100 grams of this food at all sessions depending on which condition they are randomized into. The chips provided to participants in each condition will be measured in grams to the tenth decimal point on an electronic food scale (Denver Instrument Co., Arvada, CO) before and after the session. The weight of the container will also be measured. Total grams of chips consumed during the session will be determined by subtracting pre- and post-consumption weight of the chips.

SECONDARY OUTCOMES:
Total grams of fruit consumed | 1 year
  The fruit used in this investigation is red grapes. Participants will be provided 100 grams or 150 grams of red grapes depending on which of the four groups they are participating in. Each individual will go through all four conditions in this investigation. Fruit provided to participants in each condition will be measured in grams to the tenth decimal point on an electronic food scale (Denver Instrument Co., Arvada, CO) before and after the session. The weight of the container will also be measured. Total grams of fruit consumed during the session will be determined by subtracting pre- and post-consumption weight of fruit.

OTHER OUTCOMES:
Relative Reinforcing Value of Foods | 1 Year
  As part of the investigation, participants will play a computer game which assesses the relative reinforcing value of the foods used. The number of points earned for each of the foods will be used to assess the relative reinforcing value of the foods.

CONTACTS AND LOCATIONS:
Overall Officials: Hollie Raynor, PhD, Principal Investigator — University of Tennessee
Locations (1):
- The University of Tennessee-Knoxville, Knoxville, Tennessee, United States